CLINICAL TRIAL: NCT06775444
Title: The Effect Of The Theory Of Planned Behavior Based Breastfeeding Education Program Given To Pregnant Women On Breastfeedıng Adaptation, Motivation, Self-Efficacy And The Tendency To Early Weaning.
Brief Title: Evaluation of the Effectiveness of a Breastfeeding Education Program Based on Planned Behavior Theory
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Aylin Tozluoğlu, MSc, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AnkaraÜ-HF-AT-01
Record Dates: First submitted 2024-12-15; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Breast Feeding
Keywords: Theory Of Planned Behavior; Breastfeeding; Self Efficacy; Motivation; Breastfeeding Adaptation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The research was planned to be conducted as a single-center, parallel group, randomized controlled experimental, prospective study in a pre-test-post-test design.
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to ensure confidentiality in the group distributions, the block randomization assignment of the intervention and control groups will be made by someone outside the research and will be received in pre-prepared opaque envelopes. A separate envelope will be prepared for each pregnant woman participating in the research and she will be asked to choose one. Pregnant women will not know which group they are in. Since the researcher will also be the implementer of the application, blinding will not be possible for the groups that the pregnant women are in. For this reason, only participant and statistician blinding will be provided in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): In addition to the routine breastfeeding training in the hospital where the study was conducted, the intervention group will be given a 2-session "Breastfeeding Education Program Based on the Theory of Planned Behavior".
  Interventions: Behavioral: Breastfeeding Education Program Based on Planned Behavior Theory
- Control group (Sham Comparator): The control group will receive routine breastfeeding training at the hospital where the study is conducted.
  Interventions: Behavioral: Routine Breastfeeding Training

INTERVENTIONS:
Behavioral: Breastfeeding Education Program Based on Planned Behavior Theory — In addition to routine breastfeeding training at the hospital where the study is conducted, the intervention group will be given a 2-session Breastfeeding Training Program Based on Planned Behavior Theory.
  Education Content:
  The importance of breast milk, the benefits of breastfeeding, the dangers of artificial feeding, putting the baby to the breast, signs of hunger in the baby, the harms of bottle and pacifier, breastfeeding positions, breast-related problems, information sources about breastfeeding, birth and breastfeeding leave for working mothers, breastfeeding in the community, the importance of environmental and professional support during breastfeeding. Insufficient milk anxiety, increasing milk intake and production, situations where milk should be expressed, milk expression methods, storage conditions of breast milk, alternative feeding methods with expressed milk, methods to be applied to increase breast milk, differences between breast milk and formula milk.
  Arms: Intervention Group
Behavioral: Routine Breastfeeding Training — The control group will receive routine breastfeeding education at the hospital where the study is conducted. Routine breastfeeding education includes the importance of breast milk and breastfeeding (benefits of breast milk and breastfeeding, correct breastfeeding technique and breastfeeding positions, time for the first feeding of the newborn, feeding method, expressing and storing breast milk, techniques for giving expressed breast milk as close as possible to breastfeeding, harms of bottle use, breast problems and coping methods). Pregnant women who give birth at the hospital where the study is conducted receive routine breastfeeding education from the breastfeeding nurse in the ward before being discharged.
  Arms: Control group

SUMMARY:
The aim of the research is to examine the effect of a breastfeeding training program based on the theory of planned behavior on Pregnant Womens' Breastfeeding Adaptation, Motivation, Self-Efficacy And The Tendency To Early Weaning.

DETAILED DESCRIPTION:
The aim of the study is to examine the effects of a breastfeeding education program based on the theory of planned behavior on breastfeeding adaptation, motivation, self-efficacy, and the tendency to stop breastfeeding.

The study was planned to be conducted as a single-center, parallel group, randomized controlled experimental, prospective study in a pretest-posttest design.

The study was planned to be conducted in the pregnancy school/breastfeeding counseling polyclinic of Düzce Atatürk State Hospital. The sample of the study will consist of pregnant women in the last trimester who meet the inclusion criteria. Considering the losses that may occur during the study process, it is planned to continue the study with a total of 88 pregnant women.

The data of the study will be collected from the patient based on the "Introductory Information Form", "Information Form Regarding Birth and Breastfeeding Process", "Breastfeeding Adaptation Scale", "Breastfeeding Motivation Scale (For Primiparous Mothers)", "Breastfeeding Motivation Scale (For Multiparous Mothers)", "Antenatal Breastfeeding Self-Efficacy Scale-Short Form", "Breastfeeding Self-Efficacy Scale-Short Form", "Breastfeeding Discontinuity Scale" and "Breastfeeding Follow-up Form".

In the study, the "Breastfeeding Education Program Based on Planned Behavior Theory" consisting of 2 sessions will be applied to the intervention group, while the routine breastfeeding education in the hospital where the study is conducted will be applied to the control group. The breastfeeding process will be followed for 6 months after birth in both groups.

In the analysis of the study, it is planned to analyze descriptive statistics (number, percentage, mean and standard deviation), significance test of the difference between two means in independent groups (t test), t test in dependent groups, multi-way and one-way variance analysis in repeated measurements, Pearson correlation analyses for the relationships between the dimensions determining the scale levels, and the chi-square homogeneity test for whether the intervention and control groups are homogeneous in terms of characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Those who are over 18 years old
* Pregnant women in their last trimester (pregnant women who are 27 weeks or more)
* Those who receive breastfeeding training at the Pregnancy School
* Speak and understand Turkish
* Do not have a risky pregnancy diagnosis
* Do not have multiple pregnancies
* Do not have a psychiatric or neurological disease that will affect their cognitive functions
* Have the WhatsApp application on their phone
* Volunteer to participate in the research
* Want to breastfeed their baby
* Have given birth at >37 weeks of pregnancy
* Have a baby weighing at least 2500 grams
* Have a single healthy baby in the postpartum period
* Mothers who do not have breast problems that prevent breastfeeding, do not use medication that passes into breast milk, or have any disease (such as active tuberculosis, HIV) were determined as follows.

Exclusion Criteria:

* Those who could not continue the study for any reason
* Those who did not participate in all final tests
* Those who did not participate in all training
* Those who could not be reached more than 5 times in each planned telephone/face-to-face meeting.
* Those whose babies were hospitalized in neonatal intensive care after birth (except for babies hospitalized for more than 24 hours - due to neonatal jaundice)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Attrition Prediction Tool (BAPT) | Pre-test application after routine breastfeeding education, Post-test application after the Breastfeeding Education Program Based on Planned Behavior Theory, 7-14 days postpartum, 4-6 weeks postpartum, 4th month postpartum, Postpartum 6th month
  Breastfeeding Attrition Prediction Tool (BAPT) is a scale consisting of 90 questions on a 5-point Likert-type scale based on the theory of planned behavior. There are four different sub-dimensions in the scale, which does not have a total score. These are "Negative Breastfeeding Attitude", "Positive Breastfeeding Attitude", "Social and Professional Support" and "Breastfeeding Control" and each sub-scale is scored separately. A high scale score indicates that the mother has high breastfeeding control.

SECONDARY OUTCOMES:
Breastfeeding Self-Efficacy Scale Short Form (Antenatal Breastfeeding Self-Efficacy Scale) | 1. A pre-test will be applied before the Breastfeeding Education Program Based on Planned Behavior Theory. 2. Postpartum 7-14 days 3. Postpartum 4-6 weeks 4. Postpartum 4th month 5. Postpartum 6th month
  A 14-item short form of the Breastfeeding Self-Efficacy Scale was created. He stated that the short version of the Breastfeeding Self-Efficacy Scale could also be used during pregnancy by using the phrase "future tense" in its items. The short form of the scale provides ease of application and accurately evaluates self-efficacy. Cronbach's alpha value of the scale was found to be 0.94. The scale was created on a five-point Likert type, where 1 = not at all sure and 5 = always sure. A minimum of 14 and a maximum of 70 points can be obtained from the scale. As the score increases, it means that breastfeeding self-efficacy increases
Breastfeeding Adaptation Scale (BFAS) | 7-14 days postpartum
  The 27-item scale evaluates breastfeeding adaptation. It has 8 sub-dimensions: emotional change between the mother and her baby (4 items), breastfeeding confidence (5 items), sufficient breast milk (3 items), baby's nutritional capacity and growth (4 items), familiarity with the baby (4 items), discomfort during breastfeeding (3 items), preservation of breast milk volume (2 items) and receiving social support (2 items). It was developed on a 5-point Likert type scale, where 1=Strongly agree, 5=Strongly disagree. A minimum of 27 and a maximum of 135 points can be obtained from the scale. The higher the score obtained from the scale, the higher the breastfeeding adaptation.
Breastfeeding Motivation Scale (For Primiparous Mothers) | 1.Postpartum 7-14 days, 2. Postpartum 4-6 weeks, 3. Postpartum 4th month, 4. Postpartum 6th month
  Breastfeeding motivation scale (For primiparous mothers) consists of 5 sub-dimensions and 23 items. Scale items are graded from 1=I strongly disagree to 4=I strongly agree. The scale is a 4-point Likert type, and each item is scored between 1-4. There is no total score for the scale. The scores of the sub-dimensions are calculated by taking the average of the scale sub-dimension scores. As the score obtained from the scale sub-dimension increases, the motivation representing that sub-dimension also increases. The Cronbach Alpha coefficient of the scale is 0.88.
Breastfeeding Motivation Scale (For Multiparous Mothers) | 1.Postpartum 7-14 days, 2. Postpartum 4-6 weeks, 3. Postpartum 4th month, 4. Postpartum 6th month
  Breastfeeding motivation scale (For Multiparous Mothers) consists of 6 sub-dimensions and 24 items. The Cronbach alpha value of the scale is 0.914. Scale items are graded from 1=I strongly disagree to 4=I strongly agree. The scale is a 4-point Likert type, and each item is scored between 1-4. There is no total score for the scale. The scores of the sub-dimensions are calculated by taking the average of the scale sub-dimension scores. As the score obtained from the scale sub-dimension increases, the motivation representing that sub-dimension also increases.
Breastfeeding Tracking Form | 1. The first 48 hours after birth, 2.Postpartum 7-14 days, 3. Postpartum 4-6 weeks, 4. Postpartum 4th month, 5. Postpartum 6th month
  The "Breastfeeding Tracking Form" includes the baby's feeding style, breastfeeding frequency, giving additional food other than breast milk, problems with breastfeeding, desire to continue breastfeeding, doctor's evaluation of the baby's weight gain, daily urine amount, and a chart for tracking pacifier and bottle use in order to track the breastfeeding process after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Başak Demirtaş, Principal Investigator — Ankara University Faculty of Nursing Department of Nursing; Aylin Tozluoğlu, Study Chair — Ankara University Health Sciences Institute PhD student

IPD SHARING:
Plan to Share IPD: No